CLINICAL TRIAL: NCT02084095
Title: The Role of Insulin-like Growth Factor-I (IGF-I) and Free Fatty Acids in Insulin Resistance, Insulin Secretion and Glucose Metabolism Abnormalities in Acromegaly
Brief Title: IGF-I and Free Fatty Acids Isn Glucose Metabolism in Acromegaly
Status: Completed | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Dan Niculescu, Assistant Lecturer, PhD, Carol Davila University of Medicine and Pharmacy
Other Study IDs: 28332
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background Glucose metabolism abnormalities are frequent in acromegaly. Insulin resistance (IR) correlates with the intensity of acromegaly and Insulin-like Growth factor-I (IGF-I) correlates better with IR than growth hormone (GH). Insulin secretion (IS) is significantly reduced in hyperglycemic acromegalics as compared with those with normal glucose levels. IS is independent of acromegaly intensity.

The aim of this study is to show that in active acromegaly: 1) IGF-I does not cause IR but is just a better marker of acromegaly intensity than GH; 2) high GH levels induce IR through free fatty acids (FFA); 3) hyperglycemia is caused by a defficient IS on a background of IR.

Methods Intensity of acromegaly will be assessed using serum levels of GH, IGF-I and IGF binding globulin-3. IR and IS will be assessd using an intravenous glucose tolerance test acording to Bergman model. FFA will be directly measured in plasma.

ELIGIBILITY:
Inclusion Criteria:

* active acromegaly based on following criteria: minimum GH in oral glucose tolerance test (OGTT) over 1 ng/mL and serum IGF-I over upper limit of normal for age and sex
* age between 18 and 65 years old

Exclusion Criteria:

* more than one previous pituitary surgical intervention for acromegaly
* present medical treatment for acromegaly (somatostatin analogs, GH-receptor blockers, dopaminergic agonists)
* previous pituitary radiotherapy
* present medical treatment for hyperglycemia (oral antidiabetic drugs, insulin, etc)
* pituitary failure, treated or not
* medical or surgical conditions which, in the oppinion of the principal investigator, could impact on study results or patient's safety
* fasting blood glucose over 200 mg/dL or HbA1c over 8%.
* body mass index less than 20 or over 35 kg/mp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will prospectively include patients with active acromegaly assessed in a tertiary center. All patients who meet inclusion and exclusion criteria will be invited consecutively to participate in the study until the proposed number of patients is reached.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
The correlation coefficient between IGFBP-3 and insulin resistance assessed using Bergman model is non-inferior to the correlation coefficient between IGF-I and insulin resistance | 2 years
Free fatty acids correlates significantly with insulin resistance assessed using Bergman model | 2 years
Disposition index calculated using Bergman model is significantly reduced in subjects with glucose intolerance than in subjects with normal glucose tolerance | 2 years

SECONDARY OUTCOMES:
GH, IGF-I and IGFBP-3 significantly correlates with insulin resistance calculated using Bergman model | 2 years
GH, IGF-I and IGFBP-3 significantly correlates with free fatty acids | 2 years
GH, IGF-I and IGFBP-3 does not correlate with insulin sensitivity calculated using Bergman model | 2 years
GH, IGF-I and IGFBP-3 does not correlate with disposition index | 2 years
Disposition index after reduction of acromegaly activity by various treatments | 3 months after surgery or start of medical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- "C. I. Parhon" Institute of Endocrinology, Bucharest, Romania